CLINICAL TRIAL: NCT04137198
Title: The Effect of Intranasal Sufentanil on Acute Posttraumatic Pain. A Randomized Study.
Brief Title: Sufentanil Intranasal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUFIN002
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Emergencies; Pain, Acute; Analgesia; Sufentanil
Keywords: emergency; pain; analgesia; intranasal; sufentanil
MeSH Terms: conditions — Emergencies; Acute Pain; Agnosia; Pain | interventions — Sufentanil

STUDY DESIGN:
Intervention Model Description: randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): classic analgetic protocol
- intervention (Experimental): intranasal Sufentanil
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — intranasal administration of Sufentanil Forte 0,5mcg/kg as first dose and 0,3mcg/kg as titration doses
  Other Names: Sufenta Forte
  Arms: intervention

SUMMARY:
Study of the effects of intranasal sufentanil on patients presenting to the emergency department with acute post-traumatic pain.

DETAILED DESCRIPTION:
In this study, patients presenting to the emergency department with post-traumatic pain of 7 or more on the visual analog pain scale, since less than 24 hours, in the limbs, spine or thorax are randomized in a control arm or an interventional arm.

The patients in the control arm will receive the institution's classical analgetic protocol level 1 and 3, the patients in the intervention arm are given classical level 1 medication as well as intranasal Sufentanil.

Pain is then measured using the Visual Analogue Pail Scale at 15-20 minutes and at 60 minutes. At both these time points, adverse effects and vitals are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* posttraumatic pain + lasting for less than 24 hours + with an analog visual pain scale of 7/10 or more

Exclusion Criteria:

* pregnant
* <18 years
* prisoners
* lesions of head, face or abdomen
* no consent given or possible
* pain not scorable
* known drug abuse or substitution therapy
* chronic level 3 pain medication
* intake of level 3 < 8 hours
* intoxicated patient
* allergy or intolerance to opiates
* renal or hepatic insufficiency
* < 50kg body weight
* hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
change in pain score | 15-20 minutes after first administration of Sufentanil
  pain score is measured using an analogue visual pain reporting scale (0-10, 0 for no pain at all and 10 for worst pain imaginable)

SECONDARY OUTCOMES:
change in pain score | 60 minutes after first administration of Sufentanil
  pain score is measured using an analogue visual pain reporting scale (0-10, 0 for no pain at all and 10 for worst pain imaginable)

OTHER OUTCOMES:
number of participants with adverse effects | at 15-20 and at 60 minutes
  subjects are questioned and examined for known adverse effects of Sufentanil

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
After publication all IPD will be made available through researchgate.com profile of backup investigator
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
Access Criteria: access will be granted to any researcher requesting access through Researchgate.com

REFERENCES:
- [Derived] Malinverni S, Kreps B, Lucaccioni T, Bouazza FZ, Bartiaux M, Plumacker A, Pascu A, Youatou Towo P. Effect of intranasal sufentanil on acute post-traumatic pain in the emergency department: a randomised controlled trial. Emerg Med J. 2024 Jan 22;41(2):83-88. doi: 10.1136/emermed-2023-213353. PMID 37770120